CLINICAL TRIAL: NCT02996578
Title: Consumption of Polyphenol Rich Cocoa Products Over 8 Weeks and Its Effect on Cognitive Function in Individuals in Their 5th Decade of Life.
Brief Title: Effect of Polyphenol-rich Cocoa Products on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Ruth Ashaye, Principal Investigator, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QueenMUra
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Healthy Ageing
Keywords: Cognition; Cacao; Flavan-3-ols; Blood Pressure; hemoglobin A1c protein, human; Memory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solid Matrix - Intervention (Active Comparator): Dietary Supplement: polyphenol rich chocolate bar
  17.5g of commercially available dark chocolate will be consumed daily for 8 weeks
  Interventions: Dietary Supplement: polyphenol rich chocolate bar
- Powder Matrix - Intervention (Active Comparator): Dietary Supplement: polyphenol rich cocoa powder
  6g of commercially available cocoa powder (provided as 6 x 1g gelatine capsules) will be consumed daily for 8 weeks
  Interventions: Dietary Supplement: polyphenol rich cocoa powder
- Solid Matrix Intervention - Placebo (Placebo Comparator): Dietary Supplement: low polyphenol chocolate
  17.5g of commercially available, nutritionally similar, dark chocolate will be consumed daily for 8 weeks
  Interventions: Dietary Supplement: low polyphenol content chocolate bar
- Powder Matrix - Placebo (Placebo Comparator): Dietary Supplement: nutritionally similar low polyphenol cocoa powder
  6g of commercially available, nutritionally similar, cocoa powder (provided as 6 x 1g gelatine capsules) will be consumed daily for 8 weeks
  Interventions: Dietary Supplement: low polyphenol content cocoa powder

INTERVENTIONS:
Dietary Supplement: polyphenol rich chocolate bar — High polyphenol content chocolate bar. Each participant will consume 581.4mg of polyphenols
  Arms: Solid Matrix - Intervention
Dietary Supplement: polyphenol rich cocoa powder — High polyphenol content cocoa powder. Each participant will consume 6g containing 554mg of polyphenols
  Arms: Powder Matrix - Intervention
Dietary Supplement: low polyphenol content chocolate bar — Low polyphenol content matched chocolate bar. Each participant will consume 198.5mg of polyphenols
  Arms: Solid Matrix Intervention - Placebo
Dietary Supplement: low polyphenol content cocoa powder — Low polyphenol content cocoa powder. Each participant will consume 6g containing 191.2mg of polyphenols
  Arms: Powder Matrix - Placebo

SUMMARY:
This project aims to investigate whether consumption of cocoa polyphenols has an impact on cognitive function in individuals aged 50 to 60 years of age and if such an improvement is a result of an improvement in risk factors associated with cognitive decline in ageing.

DETAILED DESCRIPTION:
Healthy cognitive ageing is an important aspect of the ageing process as it involves larger numbers of people compared to those who have already been diagnosed with conditions on the dementia spectrum (Deary et al, 2009). Hence, an active effort looking at potential lifestyle factor modification interventions to help maintain cognitive well-being are warranted.

With an ageing population, the prevalence of cognitive syndromes such as Alzheimer's disease and Parkinson's disease increases (Vauzour, 2012). Nutritional interventions can play a role in successful ageing by helping to delay the onset of age-related conditions (Hendrickx, McEwen & van der Ouderaa, 2005; Brown, Riby & Reay, 2009; Monti, Moulton & Cohen, 2015). Studies have investigated the potential role of polyphenols as part of a neuroprotective lifestyle. Mouse model studies have looked at varying polyphenol sources such as tea (Haque et al., 2006; Kaur et al., 2008), blueberry (Shukitt-Hale et al., 2015; Williams et al., 2008), Gingko Biloba (Shif et al., 2008) and cocoa (Bisson et al., 2008) to mention a few.

Ageing and neurodegenerative diseases are caused by neuronal death which in turn can be triggered by neurotoxins, neuroinflammation and specific genetic mutations (Bishop, Lu & Yankner, 2010). Dietary polyphenols have been observed to provide neuroprotection against cellular alteration by modulating the neuronal function against endogenous neurotoxins and inhibition of glial induced neuroinflammation (Vauzour, 2012).

ELIGIBILITY:
Inclusion Criteria:

* Males & Females aged 50-60years of age with normal or corrected to normal vision
* BMI cut off points of ≥18.5 to ≤29.9 kg/m2
* Waist circumference smaller than 102cm for males & smaller than 88cm for women
* Blood pressure of ≥ 90 over 60 and ≤ 120 over 80
* MoCA test score ≥ 26

Exclusion Criteria:

* Allergies to cocoa or any other ingredients commonly found in cocoa confectionary eg: milk, nuts, soya
* Smoker
* Women who are new or expecting mothers, maybe or are currently pregnant and/or breastfeeding
* Taking medications for chronic conditions including (but not limited to) diabetes, heart disease, hypertension
* No previous history of stroke, brain trauma and other head-related injuries
* No diagnosis of depression and/or anxiety
* No previous cancer diagnosis
* Taking antibiotics
* Taking steroids and non-steroidal anti-inflammatory drugs (NSAIDS)
* Women on Hormone Replacement Therapy (HRT)
* Taking medication that can cause drowsiness or affect cognitive functioning
* Taking polyphenol supplements including (but not limited to) green tea extract, acai berry extract
* Taking soy/a supplements
* History of alcohol misuse
* Fear of needles and/or fainting when blood is taken

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | 8 weeks
  A test battery consisting of 7 tests will be used to investigate the role of cocoa flavanols on cognitive function in the cohort.

SECONDARY OUTCOMES:
Blood Pressure | 8 weeks
Pulse Wave Analysis | 8 weeks
  Carotid to femoral Pulse Wave Velocity (PWV) and Augmentation Index (Aix) will be measured using a Vicorder.
Glycated Haemoglobin (HbA1c) | 8 weeks
Weight (Kg) | 8 weeks
  To allow for BMI measurement
Height (m) | 8 weeks
  To allow for BMI measurement
Body Fat Percentage | 8 weeks
Energy intakes (Kj) | 8 weeks
Flavonoid intakes (mg) | 8 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Margaret University, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deary IJ, Corley J, Gow AJ, Harris SE, Houlihan LM, Marioni RE, Penke L, Rafnsson SB, Starr JM. Age-associated cognitive decline. Br Med Bull. 2009;92:135-52. doi: 10.1093/bmb/ldp033. PMID 19776035
- [Background] Vauzour D. Dietary polyphenols as modulators of brain functions: biological actions and molecular mechanisms underpinning their beneficial effects. Oxid Med Cell Longev. 2012;2012:914273. doi: 10.1155/2012/914273. Epub 2012 Jun 3. PMID 22701758
- [Background] Hendrickx H, McEwen BS, Ouderaa Fv. Metabolism, mood and cognition in aging: the importance of lifestyle and dietary intervention. Neurobiol Aging. 2005 Dec;26 Suppl 1:1-5. doi: 10.1016/j.neurobiolaging.2005.10.005. Epub 2005 Nov 14. PMID 16290269
- [Background] Brown LA, Riby LM, Reay JL. Supplementing cognitive aging: a selective review of the effects of ginkgo biloba and a number of everyday nutritional substances. Exp Aging Res. 2010 Jan-Mar;36(1):105-22. doi: 10.1080/03610730903417960. PMID 20054730
- [Background] Monti JM, Moulton CJ, Cohen NJ. The role of nutrition on cognition and brain health in ageing: a targeted approach. Nutr Res Rev. 2015 Dec;28(2):167-180. doi: 10.1017/S0954422415000141. PMID 26650244
- [Background] Haque AM, Hashimoto M, Katakura M, Tanabe Y, Hara Y, Shido O. Long-term administration of green tea catechins improves spatial cognition learning ability in rats. J Nutr. 2006 Apr;136(4):1043-7. doi: 10.1093/jn/136.4.1043. PMID 16549472
- [Background] Kaur T, Pathak CM, Pandhi P, Khanduja KL. Effects of green tea extract on learning, memory, behavior and acetylcholinesterase activity in young and old male rats. Brain Cogn. 2008 Jun;67(1):25-30. doi: 10.1016/j.bandc.2007.10.003. Epub 2007 Dec 19. PMID 18078701
- [Background] Shukitt-Hale B, Bielinski DF, Lau FC, Willis LM, Carey AN, Joseph JA. The beneficial effects of berries on cognition, motor behaviour and neuronal function in ageing. Br J Nutr. 2015 Nov 28;114(10):1542-9. doi: 10.1017/S0007114515003451. Epub 2015 Sep 22. PMID 26392037
- [Background] Williams CM, El Mohsen MA, Vauzour D, Rendeiro C, Butler LT, Ellis JA, Whiteman M, Spencer JP. Blueberry-induced changes in spatial working memory correlate with changes in hippocampal CREB phosphorylation and brain-derived neurotrophic factor (BDNF) levels. Free Radic Biol Med. 2008 Aug 1;45(3):295-305. doi: 10.1016/j.freeradbiomed.2008.04.008. Epub 2008 May 5. PMID 18457678
- [Background] Shif O, Gillette K, Damkaoutis CM, Carrano C, Robbins SJ, Hoffman JR. Effects of Ginkgo biloba administered after spatial learning on water maze and radial arm maze performance in young adult rats. Pharmacol Biochem Behav. 2006 May;84(1):17-25. doi: 10.1016/j.pbb.2006.04.003. Epub 2006 Jun 5. PMID 16740301
- [Background] Bisson JF, Nejdi A, Rozan P, Hidalgo S, Lalonde R, Messaoudi M. Effects of long-term administration of a cocoa polyphenolic extract (Acticoa powder) on cognitive performances in aged rats. Br J Nutr. 2008 Jul;100(1):94-101. doi: 10.1017/S0007114507886375. Epub 2008 Jan 8. PMID 18179729
- [Background] Bishop NA, Lu T, Yankner BA. Neural mechanisms of ageing and cognitive decline. Nature. 2010 Mar 25;464(7288):529-35. doi: 10.1038/nature08983. PMID 20336135